CLINICAL TRIAL: NCT03854526
Title: Evaluation of Direct and Indirect Partial Dental Coronal Restorations Within a Dental Practice-based Research Network and a Set of Hospital-university Odontology Services
Brief Title: Evaluation of Dental Coronal Restorations
Acronym: RESTO DATA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0759
Record Dates: First submitted 2019-02-12; First posted 2019-02-26 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: History of at Least One Coronal Dental Restoration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without Gougerot Sjogren disease: New patient, or patient, with no history of a dental examination in the last six months and with at least one tooth with coronal dental restoration
  Interventions: Other: Evaluation of the quality of direct and indirect partial dental coronal restorations in adults
- Patients with Gougerot Sjogren disease: New patient, or patient, with no history of a dental examination in the last six months, with at least one tooth with coronal dental restoration and presenting a Gougerot Sjogren disease
  Interventions: Other: Evaluation of the quality of direct and indirect partial dental coronal restorations in adults

INTERVENTIONS:
Other: Evaluation of the quality of direct and indirect partial dental coronal restorations in adults — The medical and dental anamnesis are registered. In addition to the medical history questionnaire, the patient completes the self-assessment questionnaire on oral health. Then, a complete and intra-oral clinical examination is performed. The collection of clinical data is done on the dentist's chair. All data are included in the e-CRF.
  All radiographic procedures will be performed according to national guidelines. If the investigator deems it clinically necessary, a panoramic X-ray will be taken and stored in the patient's HER system. Periapical radiographs (using a parallelogram technique with a radiographic film holder) will be taken for teeth with periapical radiolucency on panoramic X-ray, or with defective coronal restoration, or when the clinician needs more information for diagnosis or planning.

SUMMARY:
The purpose of this study is to provide the latest information on the oral health status of patients, the lifetime of restorations, to quantify the incidence of defects rates on inserted restorations in conservative dentistry. Moreover, the study permits to compare needs of two different patient populations depending on the place of consultation (those consulting in hospital services and those consulting in private structures) and to compare the quality of coronary fillings in patients with of Gougerot Sjogren disease and those not affected.

A minimum sample of 840 adult subjects consecutively seen at the investigator's office over a period of 33 months is expected ; 400 subjects included in private structures and 440 subjected included in university hospital services (8 to 15 patients per investigator), including at least 40 patients with Gougerot Sjogren disease (disease prevalence = 0.1%).

The investigators of these study are 46 dentists working in private dental practices or private structures of dental care spread over the " Ile-de-France " and " Rhône-Alpes Auvergne " régions and 43 dentists working in 13 french university hospital services in odontology, including two hosting one consultation for Gougerot Sjogren disease, from the ReCOL network (Recherche Clinique en Odontologie Libérale).

ELIGIBILITY:
Inclusion Criteria:

* Patient having read and signed the information letter attesting to his/her non-opposition
* Affiliated to a social security scheme
* Patient over 18 years old
* New patient in the practice or in the hospital service, that can be a classical odontalogical service or a consultation specializing in Gougerot Sjogren disease, with no history of a dental examination less than six months old, or Patient who has not consulted in the last six months
* Patient with at least one tooth with partial coronal restoration

Exclusion Criteria:

- Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with at least one dental restoration and consultant for the first time since at least six months in a private practice, or at hospital, in a classical odontological service or a consultation specializing in Gougerot Sjogren disease.
Sampling Method: Non-Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Status of coronary obturation with a simplified notation a, b or c | At day 0
  notation is based on FDI (World Dental Federation) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte GROSGOGEAT, Professor, Study Director — Hospices Civils de Lyon; Franck DECUP, Associate Professor, Study Director — Assistance Publique des Hopitaux de Paris
Locations (61):
- France (61):
  - CHU de Bordeaux, Hôpital Xavier Arnozan, Unité de médecine bucco-dentaire, Bordeaux
  - Isabelle GIRSCHIG-ALLE, Boulogne
  - CHRU de Brest, Service Odontologie consultation spécialisée, Brest
  - CHRU de Brest, Service Odontologie, Brest
  - Stéphanie MIFSUD, Brindas
  - Laurianne DUDOUIT, Caluire-et-Cuire
  - Jean-Bruno LAFRASSE, Chambéry
  - Eric ROBBIANI, Châtillon
  - CHU Estaing, Service d'Odontologie, Clermont-Ferrand
  - APHP Hôpital Louis Mourier, Colombes
  - APHP, Hopital Henri Mondor, Service de Médecine Bucco-Dentaire, Créteil
  - Selma OULADDIAF, Créteil
  - Justine LOSSI, Décines-Charpieu
  - Nicolas KAPRIELIAN, Décines-Charpieu
  - Jérôme PIEAUD, Échirolles
  - Laura COHEN BOULAKIA, Échirolles
  - Alix SAUVAGNAC, Garches
  - François-Marie DUTOUR, Issoire
  - APHP Hôpital Charles Foix, Service Odontologie consultation spécialisée, Ivry-sur-Seine
  - APHP Hôpital Charles Foix, Service Odontologie, Ivry-sur-Seine
  - Camille TOURNADRE, La Fouillouse
  - Aurélie TRUFFINET, Le Mesnil-Saint-Denis
  - CHU Lille, Service d'Odontologie, Lille
  - Valentin GARYGA, Lyon
  - Marie-Anne MY, Lyon
  - Stéphanie GAUTHEROT, Lyon
  - Alexandra DAVID, Lyon
  - Arnaud JANIN, Lyon
  - Hospices Civils de Lyon, Service d'Odontologie, Lyon
  - Philippe GERENTES, Lyon
  - Jérémie DECHAUX, Montalieu
  - Claire FRANCHI, Neuilly-sur-Seine
  - Solène MARNIQUET, Neuilly-sur-Seine
  - CHU, Service d'Odontologie, Nice
  - Céline VINTER, Paris
  - Valérie AMZALLAG GUIDONI, Paris
  - Jonathan CHESNEAU, Paris
  - Anne Claire LOISEAU, Paris
  - Thibault DROUHET, Paris
  - AP-HP, Hopital Rothschlid, Paris
  - Aurélia GUERRIERI, Paris
  - Florent TREVELO, Paris
  - Christian MOUSSALLY, Paris
  - Anthony ATLAN, Paris
  - Franck DECUP, Paris
  - Magali RENEAU, Paris
  - Maxime DROSSART, Paris
  - Catherine MESGOUEZ-MENEZ, Paris
  - CHU de Reims, Pôle de Médecine Bucco-Dentaire, Reims
  - CHU, Centre de soins Dentaires, Rennes
  - Florian POCHELU, Roanne
  - Nathalie DELARGE DIONIS, Rueil-Malmaison
  - Gaëlle CHOMETTE, Saint-Just-Saint-Rambert
  - Nicolas PERIER, Saint-Marcellin-en-Forez
  - Jacques TIXIER, Solaize
  - CHU de Toulouse, Service d'Odontologie, Toulouse
  - Laure DECHELETTE, Versailles
  - Anaïs CHABANNE, Vienne
  - Harmik MINASSIAN, Villefranche-sur-Saône
  - Xavier BONDIL, Villefranche-sur-Saône
  - Nathalie JANISSET-MASSE, Villiers-sur-Marne

IPD SHARING:
Plan to Share IPD: No